CLINICAL TRIAL: NCT03192631
Title: Financial Incentives to Improve Acceptance and Adherence to Depot Injection Anti-psychotic Medication in Treatment Avoidant and Non-adherent Patients - a Pilot Study
Brief Title: Financial Incentives to Improve Acceptance of Antipsychotic Injections
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Focus Community Mental Health Team (Other)
Responsible Party: Principal Investigator, Samuel Law, Staff Psychiatrist, Focus Community Mental Health Team
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: #SMH-17-009
Record Dates: First submitted 2017-06-15; First posted 2017-06-20 (Actual); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Schizophrenia; Schizo Affective Disorder; Bipolar I Disorder
Keywords: financial incentive
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Intervention Model Description: Cross-over study of 20 patients randomized to two arms, 9 month before cross-over.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- with financial incentive (Experimental): Patients randomized to this arm will start with receiving the financial incentive. Cross-over after 9 months to treatment as usual.
  Interventions: Other: Financial incentive
- treatment as usual (No Intervention): Patients randomized to this arm will start with receiving treatment as usual, cross-over after 9 months to incentive arm.

INTERVENTIONS:
Other: Financial incentive — Incentive of $15 Canadian
  Arms: with financial incentive

SUMMARY:
There is a lack of incentive approach for patients who suffer from schizophrenia yet lack the insight to accept treatment. Most existing approaches involve coercion and involuntary hospitalizations. This study will explore whether patients with poor insight and lacking in competence for treatment decisions will improve their acceptance and adherence of depot injection antipsychotic medication if a financial incentive is offered. Ethical considerations are also explored for this innovative pilot study

DETAILED DESCRIPTION:
Background: Medication adherence in patients with schizophrenia is a major challenge. For those who do come into contact with treatment services, various clinical and psychosocial approaches to improve antipsychotic medication adherence have been studied but none is very successful. People with severe psychotic illness often have poor insight into their illness, and lack competence for treatment decisions, making them very vulnerable to frequent illness relapses due to inadequate or lack of treatment. Furthermore, to compel them to receive treatment out of concerns for their own and others' safety and welfare, they are often subjected to involuntary hospitalization and community based treatments, by means such as Community Treatment Orders (CTO). Under the authority of CTO, patients need to take medication or they will be forcefully brought to the hospital for assessment and or hospitalization. There is concern for the coercive nature of these means that may harm these patients' relationship to the psychiatric system, and overall quality of life. There is well found concern for potential violation of the ethical principle of "do no harm", particularly when less coercive, easy to understand alternatives - such as financial incentives to take medication - have not been well explored. This study aims to assess financial incentive as a promoter of medication adherence in the most medication resistant patient population.

Methods: In a randomized cross-over study, the investogators will study medication adherence by focusing exclusively on a form of medication that is accurately measureable - the long-acting injectable antipsychotic medication. Participants will be recruited from the 160 patients who are currently enrolled at the St. Michael Hospital's Assertive Community Treatment team (FOCUS). Any patient who has had less than 75% adherence rate of his/her injectable antipsychotic depot medication in the last 4 months will be recruited. There are estimated 20-30 patients who would meet the inclusion criteria. Ten patients will be randomly assigned to each arm of the cross-over study. The treatment A arm would be offered the intervention of a $15 incentive to take the injectable medication. The treatment B arm would be treatment as usual as per FOCUS services. Each phase of the cross-over study would last 9 months - i.e. the cross-over would take place after 9 months. The primary outcome will be depot medication adherence levels, comparing the adherence rates in the treatment as usual phase. The secondary outcomes will be global clinical improvement, number of voluntary and involuntary hospital admissions and Emergency Room visits, number of police and justice system encounters, number of attempted and completed suicides, incidents of physical violence, number of days spent in work/education/rehabilitation programs, subjective quality of life and satisfaction with medication. The investigators will also study the cost effectiveness of offering financial incentives.

Discussion: The pilot study aims to provide new evidence on the effectiveness and cost effectiveness of offering financial incentives as an alternative to existing coercive approaches to improving medication adherence for patients with severe psychotic disorders. If found effective, and the benefits outweigh the risks, the potential to expand the practice, under strict ethical considerations and monitoring, at a larger policy and as an optional, available service improvement tool, is anticipated to be large. This will be the first known Canadian study on the subject.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria are the following: 1) an established psychiatric diagnosis of schizophrenia, schizoaffective disorder, or bipolar disorder according to DSM-V; 2) part of the FOCUS team for at least 4 months; 3) between 18 and 65 years of age; 4) capacity to give informed consent to participate in the study; 5) be prescribed depot antipsychotic medications more than 4 months; 6) poor adherence to anti-psychotic medication, i.e. receiving less than 75% of their prescribed depot medication in the defined period of last 4 months (some patients may eventually accept depot after repeated efforts by clinicians, but the 4-month timeframe allows precise calculation of their adherence rate); and 7) team consensus on history of failure of other general methods available to the team to ensure adherence to medication (e.g. repeated psychoeducation, case meetings, family persuasion, offering of at-home depot administration, etc.); and 8) established incapacity for treatment decision.

Exclusion Criteria:

* Exclusion criteria are: 1) established learning disorder; 2) inability to give informed consent for the study; and 3) established incapacity for treatment decision.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-07-01 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Adherence to depot injection | 18 months
  The primary outcome is adherence to depot medication during the 18-month study period. Adherence will be measured, objectively, as the percentage of prescribed depot injections actually taken.

SECONDARY OUTCOMES:
The time 'delayed' in taking depot | 18 months
  The percentage of the prescribed time interval that has elapsed before the depot is taken
Clinical status | 18 months
  As assessed on the Brief Psychiatric Rating Scale -Expanded (BPRS-E), by the treating psychiatrist.
Psychosocial status | 18 months
  As assessed by the Multnomah Community Ability Scale, by the primary clinician at the beginning and end of the study.
Number of involuntary and voluntary hospital admissions | 18 months
  Any admission during the study
Number of attempted and completed suicides | 18 months
  Tracked by team
Subjective satisfaction with medication | 18 months
  Assessed by semi-structured interview
Subjective quality of life measure | 18 months
  Assessed by semi-structured interview
Incidences of physical violence during the study | 18 months
  Tracked by team
Incidences of police arrests during the study | 18 months
  Tracked by team
Days spent incarcerated during the study | 18 months
  Tracked by team
Qualitative feedback from the teams on all aspects of their experiences with the study at the beginning and end of study | 18 months
  Conducted by researcher in focus group
Costs analyses | 18 months
  cost effectiveness study by experts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Priebe S, Burton A, Ashby D, Ashcroft R, Burns T, David A, Eldridge S, Firn M, Knapp M, McCabe R. Financial incentives to improve adherence to anti-psychotic maintenance medication in non-adherent patients - a cluster randomised controlled trial (FIAT). BMC Psychiatry. 2009 Sep 28;9:61. doi: 10.1186/1471-244X-9-61. PMID 19785727